CLINICAL TRIAL: NCT01396850
Title: THE ROLE OF BBB BREAKDOWN IN THE PATHOGENESIS OF PSYCHIATRIC DISORDERS
Brief Title: Measurments Of BBB Breakdown In The Pathogenesis Of Psychiatric Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Other Study IDs: sor497310ctil
Record Dates: First submitted 2011-07-17; First posted 2011-07-19 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Psychosis
Keywords: Psychotic Patients
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Psychotic Group
- Anxiety
- Depressed
- Control Group

SUMMARY:
BBB dysfunction has been indicated in some groups of schizophrenia patients by measuring increased albumin and immunoglobulin (IgG) cerebrospinal fluid (CSF) levels. Most of the authors described a raised protein level in 5-20% of the schizophrenic patients (Muller & Ackenheil, 1995). Increased S100B levels were demonstrated in the serum of patients suffering from schizophrenia as well as depression, and this may reflect increased BBB permeability. Furthermore, this increase remains in those patients who develop a residual state with relevant negative symptoms, whereas S100B levels normalize in recovering patients (Shalev, Serlin & Friedman, 2009). CSF albumin and CSF IgG values correlate significantly with some of the SANS (Scale for the Assessment of Negative Symptoms) subscales and the SANS total score, this shows the correlation between BBB permeability and behavioral changes. It is important to say that although negative symptoms are often signs of chronicity of the disease, the abnormal CSF findings in Muller's experiment (1995) are not related to the duration of the disease, because the patients were quite young and the duration of the disease was less than 3 years.

The investigators hypothesize that a primary vascular pathology, which leads to BBB breakdown, will result a leakage of serum-derived vascular components in to the brain tissue and may cause brain dysfunction such as disturbed thinking processes, mood and behavior, as we can see in psychiatric patients.

ELIGIBILITY:
Inclusion Criteria: Psychotic, affective disorders or anxiety disorders patients admitted to Soroka Medical Center from the psychiatric hospital or self admissions to the Psychiatric department.

Patients were evaluated by study psychiatrist. Signed informed consent by the patient or his legal custodian. Subjects Age 16-65 years.

-

Exclusion Criteria:1. Patients with neurological disease, including epilepsy, ischemic stroke, multiple sclerosis, Parkinson's disease, etc.

2. Drug or alcohol abuse. 3. Patients that will need anesthesia in order to perform the MR study (not including patients who are already ventilated).

4. Patients with metal foreign body, or other contraindication to MR (according to the MR regulations).

5. Tourists or foreign residents that long terms follow up is not feasible for them.

6. Patients with renal failure / any other kind of kidney problems. 7. Pregnant women. 8. Patient with brain-injury. 9. Suicidal patients/patients with high risk for suicide/violent patients or patients that their condition might deteriorate due to participation in this study.

-

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Psychotic, affective disorders or anxiety disorders patients admitted to Soroka Medical Center from the psychiatric hospital or self admissions to the Psychiatric department.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)